CLINICAL TRIAL: NCT05908773
Title: An Open-Label, Single-Center, Phase 0, Microdose Study to Demonstrate Delivery of TTX-MC138-NODAGA-Cu64 to Radiographically Confirmed Metastases in Subjects With Advanced Solid Tumors
Brief Title: A Microdose Study of TTX-MC138-NODAGA-Cu64 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: TransCode Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TTX-MC138-NODAGA-Cu64-001
Record Dates: First submitted 2023-05-26; First posted 2023-06-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: TTX-MC138-NODAGA-Cu64 — TTX-MC138-NODAGA-Cu64 solution was developed as a PET radiopharmaceutical to permit assessment of delivery of TMX-MC138 to metastatic lesions in subjects with solid tumors. Subjects will be administered a microdose of TTX-MC138-NODAGA-Cu64 injection administered intravenously followed by whole body PET imaging.

SUMMARY:
This is an open-label, single-center, single-arm, phase 0, microdose study in subjects with advanced solid tumors and radiographically confirmed metastases.

The study will evaluate delivery of TTX-MC138-NODAGA-Cu64 radiographically and establish the PK and biodistribution of TTX-MC138-NODAGA-Cu64 as determined by PET-MRI. The study consists of 3 parts: a screening period, dosing period, and follow-up period. The estimated total duration of the study is approximately 46 days.

Approximately 12 subjects with advanced metastatic solid tumors will be enrolled at 1 single site.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent form for the study prior to the performance of any study-specific procedures.
2. Greater than or equal to 18 years of age at the time of screening.
3. Histologically or cytologically confirmed diagnosis of metastatic solid tumor that is not amenable to curative therapy unless participation in the study would delay standard therapy.
4. Eastern Cooperative Oncology Group performance status of 0 to 1.
5. Adequate organ function defined as:

   1. Platelet count ≥100 × 109/L with no platelet transfusions in the past 7 days
   2. Absolute neutrophil count ≥1.5 × 109/L
   3. Hemoglobin ≥9 g/dL (red blood cell transfusion may be used to reach 9 g/dL but must have been administered at least 1 week prior to the administration of the study drug)
   4. Aspartate aminotransferase or alanine aminotransferase <3 × the upper limit of normal (ULN) if no hepatic metastases are present; <5 × ULN if hepatic metastases are present
   5. Total bilirubin <1.5 × ULN; <3 × ULN in the presence of Gilbert's disease
   6. Estimated (Cockcroft-Gault formula) or measured creatinine clearance ≥50 mL/min
6. At least 1 target lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (at least 10 mm per MRI from fludeoxyglucose [FDG] PET-MRI).
7. Women of childbearing potential must either abstain from sexual intercourse or employ highly effective contraception measures during the study and for at least 30 days after the administration of the study drug. Highly effective measures include 2 forms of contraception. Postmenopausal or surgically sterile women (ie, hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) are eligible. Postmenopausal status is defined as either: amenorrheic for ≥12 months following cessation of exogenous hormonal treatments and without an alternative medical cause; luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for women under 50 years of age; radiation-induced ovarian ablation with last menses ≥1 year ago; or chemotherapy-induced menopause with a ≥1-year interval since last menses. Female subjects must refrain from donating or banking eggs (ova, oocytes) and retrieving eggs for use during study treatment and for 30 days after the administration of the study drug.
8. Male subjects, if not surgically sterile, must either abstain from sexual intercourse or employ highly effective contraception (condoms or other barrier forms of contraception) during the study and for at least 30 days after the administration of the study drug. Male subjects should also avoid semen donation or providing semen for in vitro fertilization during the above-mentioned duration.
9. If a clinically indicated MRI is planned, it must be completed at least two weeks prior to or at least two weeks post investigational drug administration.

Exclusion Criteria:

1. Unwilling or unable to comply with scheduled visits, study drug administration plan, laboratory tests, or other study procedures and study restrictions.
2. QT interval corrected using Fridericia's formula >480 ms. Subject has a history of prolonged QT syndrome or torsade de pointes. Subject has a familial history of prolonged QT syndrome.
3. Clinically significant, uncontrolled cardiovascular disease including congestive heart failure class III or class IV according to the New York Heart Association classification; myocardial infarction or unstable angina within the previous 6 months; uncontrolled hypertension (Grade 3 or higher); or clinically significant, uncontrolled arrhythmia, including bradyarrhythmias that may cause QT prolongation (eg, type II second-degree heart block or third-degree heart block).
4. Symptomatic central nervous system (CNS) metastases or primary CNS tumor that is associated with progressive neurologic symptoms or requires ongoing corticosteroids to control the CNS disease. Subject must have a stable neurologic status without steroid support for at least 2 weeks before the start of study drug administration. Subjects with stable or asymptomatic CNS metastases or primary CNS are eligible. Brain computed tomography/MRI with or without contrast is mandatory within 4 weeks before the start of study drug administration in case of clinical evidence of brain metastatic disease.
5. Subject who has received anticancer therapy (including both systemic therapy and radiotherapy, but not including immunotherapy or other antibody therapies) within 14 days or 5 half-lives (whichever is shorter) of study drug administration or received antibody therapy within 28 days before the start of study drug administration. The study drug may be started within these washout periods if considered by the investigator to be safe, except on the day of study drug administration.
6. Prior radiation therapy is allowed, provided >14 days have elapsed since completion of radiation prior to enrollment. If target lesions were radiated, they should have progressed prior to the administration of the study drug to be considered target lesions per Response Evaluation Criteria in Solid Tumors version 1.1. If the prior radiation exposure in research studies in the previous 12 months exceeds the current guidelines (ie, 50 mSv/year), the subject will not be enrolled.
7. Administered a radioisotope within 10 physical half-lives before the start of study drug administration.
8. Subject is unable to undergo or has a contraindication to PET or MRI scan.

   * Subject who has electrical implants such as cardiac pacemaker or perfusion pump
   * Subject who has claustrophobic reactions
   * Body weight over the weight limit for the moving table (>300 lbs for the MRI)
   * Unable to lie comfortably on a bed inside the PET scanner
   * Metallic or electric implants contraindicated for PET-MRI scanning when applicable
9. Subject who has an advanced solid tumor with metastasis to liver only, lymph nodes only, or liver and lymph nodes only.
10. Subject who requires treatment with traditional/herbal medicines or their preparations indicated for tumors or with adjuvant antitumor effects that cannot be discontinued for the day of study drug administration.
11. Subject who received a major surgical procedure within 28 days before the start of study drug administration (procedures such as central venous catheter placement and tumor needle biopsy are not considered major surgical procedures). The study center should discuss other minor surgeries with the sponsor.
12. History of another primary malignancy that has been diagnosed or required therapy within the past year. Note: The following prior malignancies are not exclusionary: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate or breast cancer, curatively treated localized thyroid cancer, and completely resected carcinoma in situ of any site.
13. Subject is pregnant at the time of screening or on Day 1 before the PET-MRI, as documented by a serum beta human chorionic gonadotropin pregnancy test consistent with pregnancy.
14. Subject is breastfeeding at the time of screening.
15. Known human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus infection that meets the following criteria:

    1. Subject with HIV infection is eligible if: documented with undetectable HIV RNA within 4 weeks of study drug administration,
    2. No acquired immunodeficiency syndrome defining opportunistic infections within the past 12 months prior to study enrollment, and
    3. Is on antiretroviral therapy for at least 4 weeks prior to study enrollment.
16. Presence of any severe or uncontrolled systemic disease or condition, including: (i) uncontrolled hypertension or diabetes; (ii) serious cardiac, pulmonary, or renal conditions; (iii) active bleeding diatheses; (iv) any active type of bacterial, viral, fungal, or other infection that would pose a significant risk to the subject in the opinion of the investigator.
17. Subject who has clinical signs or symptoms consistent with COVID-19 infection or confirmed infection by appropriate laboratory test (done at the discretion of investigator or per local regulation) within the last 2 weeks before the administration of the study drug. In case of confirmed COVID-19 infection before screening, documentation of resolution of infection by appropriate laboratory test is required.
18. Subject who has received or is planning to receive a COVID-19 vaccination within 2 weeks before or after the administration of the study drug. However, COVID-19 vaccinations received >2 weeks before or after the administration of the study drug are permitted.
19. Subject who has received a live or live attenuated vaccines within 30 days before the administration of the study drug.
20. Any unresolved toxicities from prior therapy, greater than CTCAE Grade 1 at the time of starting study treatment, with the exception of alopecia.
21. History of hypersensitivity to active or inactive excipients of the study drug or drugs with a similar chemical structure or class to the study drug, including ferumoxytol (Feraheme).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Injected Dose | Throughout study completion for 12 subjects, average 12 months
  Measure the percent injected dose per cubic centimeter (%ID/cc) tissue of TTX-MC138-NODAGA-Cu64 in radiographically confirmed metastatic lesions in subjects with advanced solid tumors using PET-MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States